CLINICAL TRIAL: NCT05182138
Title: Do Zinc Fortified Potatoes Improve Zinc and Health Status?
Brief Title: Zinc in Potatoes Study
Acronym: ZIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: Fight for Sight (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02/033/15
Record Dates: First submitted 2021-12-15; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: No Conditions

STUDY DESIGN:
Intervention Model Description: 3 arms in parallel
Who Masked: Participant, Care Provider, Investigator
Masking Description: Computer-based randomisation system
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unfortified potato plus placebo (Placebo Comparator): Volunteers given potato with no fortified zinc and a placebo
  Interventions: Other: Unfortified potato plus placebo
- Zinc Biofortified potato plus placebo (Active Comparator): Volunteers given potato biofortified with zinc and a placebo
  Interventions: Other: Zinc Biofortified potato plus placebo
- Unfortified potato plus zinc supplement (Active Comparator): Volunteers given potato with no fortified zinc and a zinc supplement
  Interventions: Other: Unfortified potato plus zinc supplement

INTERVENTIONS:
Other: Unfortified potato plus placebo — Volunteers will be given 300g of zinc unfortified cooked potato as well as a placebo every day.
  Arms: Unfortified potato plus placebo
Other: Zinc Biofortified potato plus placebo — Volunteers will be given 300g of cooked potato biofortified with zinc and a placebo every day.
  Arms: Zinc Biofortified potato plus placebo
Other: Unfortified potato plus zinc supplement — Volunteers will be given 300g of zinc unfortified cooked potato and a zinc supplement containing 18mg of zinc, every day.
  Arms: Unfortified potato plus zinc supplement

SUMMARY:
Zinc is important in biology and allows the proper function of proteins in living organisms. Severe zinc deficiency in animals and humans over long periods of time can therefore cause adverse effects. In the UK, the zinc status of most people is adequate, but about 20% of the population, especially adolescents in deprived communities and vegetarians/vegans, are likely marginally zinc deficient. Because potatoes are a favoured food in adolescents and vegetarians/vegans, the investigators have improved the zinc content of Saxon potatoes by biofortification, which involves spraying potato plant leaves with zinc salts. The potato zinc concentration is about three times the level in unfortified potatoes of the same variety. This level of zinc can boost the zinc intake of people who are marginally zinc deficient so that they become zinc adequate. Indeed, in rat studies, the investigators have shown that addition of some zinc-biofortified potato to a low zinc diet improves the zinc and health status of the animals. In the present study, the investigators propose to investigate whether the potato biofortification can improve the zinc and health status of volunteers. Because most of the volunteers (healthy adult men and women after the menopause) might have normal or variable zinc status at recruitment, it might not be possible to see the benefits of the potato diets and therefore, the investigators shall reduce the zinc intake of all 45 participants to 1 mg Zn/d for a period of two weeks prior to feeding 15 randomly selected individuals the biofortified potato diets (4 mg Zn/d) for two weeks. Zinc and health status will be measured by blood tests before and after zinc depletion and after feeding the potato diets. Results will be compared with data from 15 volunteers eating unfortified potato diets with a daily placebo and 15 volunteers consuming the unfortified potato diets with a zinc supplement (18 mg/d) as a positive control.

DETAILED DESCRIPTION:
There is a small but critical window of dietary zinc intake from 1 to 4 mg Zn/day over which the symptoms of long-term zinc deficiency go from acute to chronic in nature. For example, at 1 mg Zn/day intake for several months, most people will develop skin lesions, but at 4 mg Zn/day, skin lesions would be very rare. However, impaired immune response can be detected when consuming zinc up to 6 mg/day over several months. Dietary intakes of <4 mg Zn/day in developed countries is rare but can be common in developing countries.

This study has been carefully designed to test the hypothesis that consumption of zinc biofortified potatoes can rescue the zinc status and health of people who are of low zinc status and consuming diets which are borderline acutely zinc deficient. The protocol for the study includes 2 weeks of zinc deprivation at around 1 mg Zn/day dietary intake (Very Low Zinc Diet) followed by 2 weeks of a borderline acutely/chronically deficient diet of around 4-5 mg Zn/day (Low Zinc Diet). Two weeks on the Very Low Zinc Diet has been carefully and deliberately selected to cause biochemical changes due to zinc deprivation but not signs and symptoms of deficiency such as skin lesions. Less than 2 weeks is insufficient to cause the biochemical effects and more that 2 weeks risks the physical manifestation of deficiency and also non-compliance by volunteers, since the diets may be less palatable than their habitual diet. Thus all volunteers will have low zinc status at the time of starting to eat the Low Zinc Diet, and the effect of eating the biofortified potatoes in addition, which will add an extra 1 mg to the daily zinc intake, should be seen in all the zinc and health status tests that the investigators are proposing. In rat studies in which the investigators did just this kind of intervention, the biofortified potato ameliorated the effect of zinc deficiency on growth, food intake and immune function.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18 or over
* Postmenopausal females
* Healthy
* BMI 19-35

Exclusion Criteria:

* Physical or mental health problems
* Long-term medication
* Smoking
* Alcohol >20 units/week
* Health supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Plasma Zinc status | 4 weeks
  Plasma zinc levels will be measured using ICP-MS
Zinc status | 4 weeks
  The Exchangeable Zinc Pool size (EZP) will be assessed by the analysis of the Zn stable isotopes excreted in the urine by ICP-MS/MS.

SECONDARY OUTCOMES:
Eye Electrophysiology | 4 weeks
  After overnight dark adaptation using an eye patch, electroretinograms will be recorded following dilation with eye drops G. Tropicamide 1% & G. phenylephrine 2.5%) using non-invasive corneal electrodes.
Thromboelastography (efficiency of blood clotting) | 4 weeks
  The efficiency of blood clotting within participants will be assessed by collecting whole blood samples into 3.2% sodium citrate tubes and then analysing this for blood clotting parameters using thromboelastography (ROTEM). This analysis generates 4 values representing clot formation which will be assessed and compared between the different interventions: the reaction time (R), the speed of clot formation (K-value), the angle and the maximum amplitude (MA).

CONTACTS AND LOCATIONS:
Overall Officials: John H Beattie, PhD, Principal Investigator — University of Aberdeen
Locations (1):
- University of Aberdeen, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No